CLINICAL TRIAL: NCT06988904
Title: EFFECTIVENESS OF THE GROUP-BASED NUTRITION EDUCATION PROGRAMME FOR OBESITY MANAGEMENT IN BERGUEDÀ: A RANDOMISED CLINICAL TRIAL. ENERGY2MOB STUDY
Brief Title: ENERGY2MOB STUDY: OBESITY MANAGEMENT IN BERGUEDÀ
Acronym: ENERGY2MOB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Anna Ruiz Comellas, Principal Investigator, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24/303-P
Record Dates: First submitted 2025-02-08; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Mediterranean Diet; Overweight or Obese Adults; Exercise Therapy; Cardiovascular Diseases; Psychological Well Being
Keywords: obesity and overweight; primary health care; Mediterranean diet; dietary interventions
MeSH Terms: conditions — Overweight; Cardiovascular Diseases; Psychological Well-Being; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Intervention: The Energy2MOB programme will take place at three primary healthcare centres in Berguedà: Baix Berguedà (Puig-Reig CAP), Berga Centre (Berga CAP), Alt Berguedà (Guardiola de Berguedà CAP)
  The programme will include:
  * One pre-intervention visit
  * 8 weekly group sessions
  * One post-intervention visit
  * One-month telephone follow-up
  * In-person follow-ups at three and six months
  Interventions: Other: Energy2MOB
- Control group (No Intervention): The control group will continue with standard care at their usual primary healthcare centre and will only attend pre-intervention, post-intervention, and six-month follow-up visits. They will not receive group sessions or telephone follow-ups. If the Energy2MOB programme proves effective, control group participants will be invited to participate in the intervention sessions.

INTERVENTIONS:
Other: Energy2MOB — Intervention: The Energy2MOB programme will take place at three primary healthcare centres in Berguedà:
  Baix Berguedà (Puig-Reig CAP) Berga Centre (Berga CAP) Alt Berguedà (Guardiola de Berguedà CAP)
  The programme will include:
  One pre-intervention visit 8 weekly group sessions One post-intervention visit One-month telephone follow-up In-person follow-ups at three and six months
  The control group will continue with standard care at their usual primary healthcare centre and will only attend pre-intervention, post-intervention, and six-month follow-up visits. They will not receive group sessions or telephone follow-ups. If the Energy2MOB programme proves effective, control group participants will be invited to participate in the intervention sessions.
  Arms: Interventional group

SUMMARY:
Background: Obesity is a prevalent multifactorial disease worldwide and has become a significant public health concern. The latest data from the 2022 Catalonia Health Survey show that 56.2% of men and 43.7% of women are overweight or obese, and 39% of children aged 6 to 12 years have excess weight. Excess adiposity poses a health risk as it is associated with various chronic diseases such as type 2 diabetes mellitus, hypertension, and dyslipidaemia, all of which affect quality of life and increase mortality risk.

Hypothesis: The Energy2MOB obesity management programme in Berguedà is a group-based intervention incorporating nutrition education and physical activity. It aims to reduce excess body weight and the risk of chronic diseases, including type 2 diabetes mellitus, dyslipidaemia, and hypertension, through a multicomponent approach that enhances dietary habits, physical activity, and emotional eating regulation.

Objectives

* Assess the effectiveness of the Energy2MOB programme in reducing body weight by 5-10% among adults with obesity in the Berguedà health region.
* Measure lifestyle modifications, including dietary habits, physical activity, and emotional eating.

Methodology: A randomised clinical trial with two groups (control and intervention) over one year, including individuals aged 18-65 years in the Berguedà health region with overweight grade II (BMI 27-30 kg/m²) or obesity (BMI 30-40 kg/m²). Exclusion criteria include significant language barriers, previous bariatric surgery, moderate to severe cognitive impairment, and severe psychiatric disorders preventing participation in sessions. Participants must attend at least 80% of the programme.

Measurements

* Sociodemographic factors: sex, age, education level, marital status, employment status.
* Lifestyle factors: alcohol and tobacco use, dietary habits, physical activity, emotional eating, health-related quality of life.
* Anthropometric parameters: body weight, height, BMI, waist circumference.
* Blood pressure, medication use, biochemical parameters (fasting glucose, glycated haemoglobin, lipid profile, liver and kidney function markers, C-reactive protein).

Statistical Analysis: Accepting an alpha risk of 0.05 and a statistical power above 0.8 in a bilateral contrast, 68 subjects per group are required to detect a difference of at least 2.5 kg. A common standard deviation of 4.77 is assumed, with an estimated 15% dropout rate. Sample size calculations were performed using GRANMO version 8.0 (https://www.datarus.eu/ca/aplications/granmo/; consulted in November 2024).

Expected Outcomes, Applicability, and Relevance: This study aims to generate scientific evidence on the effectiveness of multicomponent group-based interventions focused on improving nutrition, physical activity, and psychological well-being in obesity and chronic disease management. It seeks to create an environment that facilitates behavioural changes, leading to weight reduction and improved quality of life. The findings will also contribute to the development of a practical guide for addressing excess weight in primary healthcare settings.

Keywords (maximum 6): Adult obesity, primary health care, group interventions, dietary interventions, multicomponent interventions, Mediterranean diet.

DETAILED DESCRIPTION:
BACKGROUND AND CURRENT STATE OF THE TOPIC Obesity is a chronic, complex, and prevalent disease worldwide, posing a significant public health concern with high socio-economic costs. The World Health Organization (WHO) defines it as an abnormal or excessive accumulation of fat that impairs health, promotes medical complications, and reduces life expectancy.

Recent studies indicate that obesity prevalence has risen in recent years and is projected to continue increasing. According to a recent study by the Carlos III Health Institute in collaboration with the Spanish Agency for Food Safety and Nutrition (AESAN) and regional health services, 55.8% of adults are overweight (63.7% of men and 48.4% of women), and 18.7% have obesity (19.3% of men and 18.0% of women). Among children and adolescents, 10.7% have obesity, and 30% are overweight. More specifically, the 2022 Catalonia Health Survey reports that half of the population aged 18-74 years has excess weight, including overweight and obesity, with 56.2% of men and 43.7% of women affected. Among children aged 6-12 years, nearly 39% have excess body weight, with 25.2% classified as overweight and 13.7% as obese.

There is no doubt that modern society fosters an obesogenic environment, promoting sedentary lifestyles and unhealthy diets dominated by processed foods. However, additional factors predispose individuals to excess weight even without exposure to these obesogenic influences. Obesity is a multifactorial disease, involving both intrinsic (non-modifiable) factors such as genetics and physiological causes and extrinsic (modifiable) factors such as environmental, psychological, social, economic, and political influences.

Physiopathologically, obesity is characterised by chronic low-grade inflammation due to adipose tissue dysfunction caused by excessive and/or abnormal fat accumulation. Excess adiposity is a major health risk as it is associated with a broad range of chronic diseases, including cardiovascular disease, type 2 diabetes mellitus, certain cancers, mental health disorders, chronic kidney disease, musculoskeletal complications, respiratory diseases, and non-alcoholic fatty liver disease (NAFLD). Addressing this issue with evidence-based solutions is urgent and a public health priority.

Expert groups, including the National Institutes of Health, WHO, the Academy of Nutrition and Dietetics, and the Spanish Society for the Study of Obesity (SEEDO), recommend a 5-10% reduction in initial body weight over six months to achieve health benefits and manage obesity-related comorbidities. Such weight loss is associated with reductions in body mass index (BMI), waist circumference, and fat mass, alongside significant improvements in glucose levels, lipid profile, and blood pressure. Consequently, obesity reduction strategies offer substantial benefits for chronic disease management, particularly type 2 diabetes mellitus, dyslipidaemia, and hypertension.

Beyond its impact on physical health, obesity also affects emotional, psychological, and social well-being. Weight-related stigma, discrimination, and bias contribute to decreased quality of life and increased obesity-related comorbidities. Current scientific evidence highlights that body weight regulation is not solely under voluntary control, as biological, genetic, and environmental factors play fundamental roles in obesity development and maintenance. Ineffective weight loss outcomes, insufficient multidisciplinary coordination, a lack of human and economic resources for obesity management, and societal misperceptions about obesity-particularly in lower socioeconomic groups-contribute to the overburdening of healthcare systems, preventing comprehensive and high-quality patient care.

Therefore, obesity treatment must adopt a holistic approach to achieve long-term health and well-being improvements. The focus should shift from mere weight reduction to sustainable lifestyle changes, including dietary modifications, increased physical activity, and psychological well-being improvements. Effective intervention requires a multidisciplinary team of specialists (e.g., dietitians-nutritionists, physicians, nurses, psychologists, and physical activity experts) working collaboratively to enhance patient health and well-being.

More specifically, interventions should promote a well-balanced diet alongside regular physical activity and behavioural therapy to sustain long-term lifestyle changes. The Mediterranean diet, a well-established cardioprotective dietary model in the region, serves as the basis for this approach. It emphasises a high intake of natural plant-based fats (extra virgin olive oil and nuts), minimally processed plant-based foods (vegetables, fruits, legumes, and whole grains), limited meat consumption (especially red and processed meats), moderate fish and egg consumption, and minimal intake of ultra-processed foods high in saturated fats, trans fats, and added sugars.

Regular physical activity and exercise are crucial in obesity treatment as they enhance weight loss, reduce abdominal fat, support weight maintenance, improve well-being, and positively impact cardiovascular risk factors. Psychological therapy plays an essential role, incorporating motivational strategies, problem-solving techniques, stimulus control, and stress reduction techniques. The COM-B behaviour change model will underpin the multicomponent group education intervention, ensuring participant motivation and engagement throughout all obesity treatment phases-critical for achieving successful outcomes.

Although several scientific studies have demonstrated the effectiveness of lifestyle modification-based group interventions, their implementation in primary healthcare settings remains limited due to a shortage of trained professionals with adequate availability. This highlights the need for resource allocation to address the issue effectively. Developing and implementing specific programmes based on a collaborative and interdisciplinary care model is crucial for successfully managing obesity and its associated health consequences. Such initiatives could improve the prevalence of cardiometabolic risk factors in affected individuals.

In 2021, the Catalan primary healthcare system incorporated dietitians-nutritionists through the Programme for the Promotion of Healthy Eating and the Prevention and Management of Diseases in Primary and Community Healthcare. These professionals focus on preventing and treating nutrition-related health issues by promoting healthy and sustainable eating habits tailored to individual conditions, risks, diseases, preferences, and socio-economic and cultural circumstances, with a particular focus on vulnerable populations. Additionally, primary healthcare introduced other roles, such as emotional well-being and community health specialists and physiotherapists, to facilitate the implementation of such programmes.

This project builds on prior obesity management interventions in primary healthcare settings, incorporating insights from past participants to refine and enhance its effectiveness. It has the potential to generate robust evidence on the effectiveness of multicomponent group-based interventions for obesity and chronic disease management in adults, providing a supportive environment that fosters sustainable behaviour change for improved patient quality of life and optimal health outcomes. If the intervention proves successful, a practical guide will be developed for broader implementation across primary healthcare centres addressing adult obesity.

HYPOTHESIS Participation in the Energy2MOB group education programme for obesity management in Berguedà will lead to a reduction in body weight among individuals with overweight or obesity. Additionally, it will improve dietary habits, physical activity levels, and emotional eating behaviour, while also supporting the management of chronic diseases such as type 2 diabetes mellitus, dyslipidaemia, and hypertension.

OBJECTIVES Primary Objectives (PO)

* PO1: To assess the effectiveness of the Energy2MOB programme in achieving a 5-10% reduction in body weight among adults with overweight or obesity in the Berguedà healthcare region.
* PO2: To determine lifestyle changes related to adherence to the Mediterranean diet, regular physical activity, and improved emotional eating regulation.

Secondary Objectives (SO)

* SO1: To evaluate changes in biochemical, anthropometric, and blood pressure parameters.
* SO2: To analyse improvements in health-related quality of life, reduction in cardiovascular risk, and better management of comorbidities (hypertension, dyslipidaemia, and diabetes mellitus).
* SO3: To examine the feasibility of implementing the programme by assessing adherence, fidelity, and participant satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Overweight (BMI 27-30 kg/m²) or obesity (BMI 30-40 kg/m²)
* Availability to attend at least 80% (6 out of 8) of the group sessions

Exclusion Criteria:

* Significant language barriers (unable to communicate in Catalan or Spanish)
* Previous bariatric surgery
* Moderate to severe cognitive impairment
* Severe psychiatric disorders preventing participation in group sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-06-07 (Estimated); Primary Completion 2026-03-07 (Estimated); Study Completion 2026-03-07 (Estimated)

PRIMARY OUTCOMES:
Body weight changed | 1 year
  Body weight changed refers to the process of losing body weight, typically through a combination of diet, exercise, and lifestyle changes. It is aimed at changing excess body fat, improving health, and achieving a healthier body composition. This changed can vary depending on the individual's goals, metabolic rate, and overall health.

SECONDARY OUTCOMES:
Body weight | 1 year
  Calibrated scale, measured with light clothing and without shoes, in kilograms
Height | 1 year
  With stadiometer, mesured in metres
Waist circumference | 1 year
  Measured at the level of the navel using a flexible measuring tape, in centimetres
BMI (Body Mass Index) | 1 year
  Weight and height will be combined to report BMI in kg/m^2
Obesity-Related Comorbidities | 1 year
  Hypertension, dyslipidaemia/hypercholesterolaemia, type 2 diabetes mellitus, Fibromyalgia, cardiovascular disease, sleep apnoea syndrome, Osteoarticular pathology, non-alcoholic fatty liver disease (NAFLD), urinary incontinence
Medication Use | 1 year
  Medication used for comorbidities associated with obesity refers to drugs prescribed to manage health conditions that often occur alongside obesity, such as type 2 diabetes, hypertension, dyslipidemia, and sleep apnea. These medications help control the symptoms and prevent further complications related to these comorbidities.
Blood Pressure (systolic and diastolic) | 1 year
  Blood pressure refers to the force exerted by circulating blood on the walls of blood vessels. It is measured in two values: systolic and diastolic.
  Systolic blood pressure is the higher number and represents the pressure in the arteries when the heart contracts and pumps blood.
  Diastolic blood pressure is the lower number and measures the pressure in the arteries when the heart is at rest between beats.
  Normal blood pressure is typically around 120/80 mmHg. Blood pressure higher than 130/80 mmHg is considered elevated or high, which can increase the risk of cardiovascular diseases, strokes, and kidney problems. Monitoring and managing blood pressure is essential for maintaining overall health, particularly in individuals with obesity or other risk factors.
Fasting plasma glucose | 1 year
  Plasma glucose refers to the concentration of glucose (sugar) in the liquid component of blood. It serves as a primary energy source for the body's cells. Measuring plasma glucose is essential for diagnosing and monitoring metabolic conditions such as diabetes mellitus. Normal fasting levels typically range between 70 and 100 mg/dL.
Glycated haemoglobin (HbA1c) | 1 year
  Glycated haemoglobin (HbA1c) reflects the average blood glucose levels over the past two to three months. It forms when glucose binds to hemoglobin in red blood cells. HbA1c is widely used to diagnose and monitor diabetes. Normal values are generally below 5.7%, with higher levels indicating poor long-term glucose control.
Smoking status | 1 year
  Current smoker, former smoker, non-smoker
Cardiovascular risk | 1 year
  Assessed using validated risk score tools, REGICOR calculator. TABLES FOR CALCULATING 10-YEAR CORONARY RISK: <5% Low risk, 5-9.9% Moderate risk, 10-14.9% High risk, ≥15% Very high risk
Mediterranean diet adherence | 1 year
  Adherence to the Mediterranean diet through the validated MEDAS questionnaire: <9 low adherence, >= 9 good adherence
Dietary habits evaluation | 1 year
  Eating behaviour questionnaire
Physical activity level | 1 year
  International Physical Activity Questionnaire (IPAQ) short version. Results:
  * Low. They do not record physical activity, or they record it but it does not meet the medium or high categories.
  * Medium. Considers the following criteria: 3 or more days of vigorous physical activity of at least 20 minutes per day. 5 or more days of moderate-intensity physical activity or walking of at least 30 minutes. 5 or more days of any combination of light, moderate, or vigorous physical activity that reach a record of 600 METs-min/week.
  * High. This is a high category and meets the following requirements: 3 or more days of vigorous physical activity or that accumulate 1,500 METs-min/week. 7 or more days of any combination of light, moderate, or vigorous physical activity that reach a record of 3,000 METs-min/week.
Emotional eating assessment | 1 year
  Emotional Eating Questionnaire (CCE) Garaulet. Scale scores: unemotional eater 0 to 5, mildly emotional eater 6 to 10, emotional eater 11 to 20, and highly emotional eater 21 to 30 points.
Health-related quality of life | 1 year
  EuroQol-5D (EQ-5D) with Visual Analogue Scale (VAS): Improvement in Health-Related Quality of Life (HRQoL) after the intervention: an improvement in HRQoL is considered if there is a decrease in the EuroQol (EQ-5D) questionnaire score compared to the baseline. A set of values consists of weights that convert each EQ-5D health profile into a value on a scale anchored between 1 (meaning complete health) and 0 (meaning a condition as serious as death).
Programme adherence | 1 year
  Based on participant attendance records
Intervention fidelity | 1 year
  Nomber of participants with completion of planned activities in each session
Programme satisfaction | 1 year
  Participant feedback survey
Total cholesterol | 1 year
  Total cholesterol measures the overall amount of cholesterol in the blood, including LDL (bad), HDL (good), and other lipid components. It is an important marker for cardiovascular health. High levels are associated with an increased risk of heart disease and stroke. Desirable values are generally below 200 mg/dL.
HDL cholesterol | 1 year
  HDL cholesterol (high-density lipoprotein) is known as the "good" cholesterol because it helps remove excess cholesterol from the bloodstream. Higher HDL levels are associated with a lower risk of cardiovascular disease. It plays a protective role in heart health. Optimal levels are typically above 60 mg/dL.
LDL cholesterol | 1 year
  LDL cholesterol (low-density lipoprotein) is often referred to as the "bad" cholesterol because high levels can lead to plaque buildup in the arteries, increasing the risk of cardiovascular disease. It is a key marker in assessing heart health. Optimal levels are typically below 100 mg/dL.
Triglycerides | 1 year
  Triglycerides are a type of fat (lipid) found in the blood, used by the body for energy. High levels can increase the risk of cardiovascular disease, especially when combined with low HDL or high LDL cholesterol. Normal fasting levels are typically below 150 mg/dL.
Alanine aminotransferase (ALT) | 1 year
  Alanine aminotransferase (ALT) is an enzyme primarily found in the liver that helps convert proteins into energy for liver cells. Elevated ALT levels in the blood may indicate liver damage or inflammation. Normal values typically range from 7 to 56 U/L.
Aspartate aminotransferase (AST) | 1 year
  Aspartate aminotransferase (AST) is an enzyme found in the liver, heart, muscles, and other tissues. It plays a role in amino acid metabolism. Elevated AST levels can indicate liver injury or damage to other organs. Normal levels usually range from 10 to 40 U/L.
Gamma-glutamyl transferase (GGT) | 1 year
  Gamma-glutamyl transferase (GGT) is an enzyme primarily found in the liver and bile ducts. It is involved in the metabolism of glutathione and the transport of amino acids. Elevated GGT levels are commonly used as a marker of liver disease, alcohol consumption, or bile duct obstruction. Normal values typically range from 0 to 30 U/L.
Creatinine | 1 year
  A waste product produced by muscles from the breakdown of creatine. It is filtered by the kidneys, and elevated levels in blood can indicate impaired kidney function.
Glomerular Filtration Rate (GFR) | 1 year
  A measure of kidney function that indicates how well the kidneys are filtering waste from the blood. It is calculated based on factors like age, sex, and creatinine levels.
C-reactive Protein (CRP) | 1 year
  A protein produced by the liver in response to inflammation. High levels of CRP in the blood can indicate inflammation or infection in the body.

CONTACTS AND LOCATIONS:
Locations (1):
- Unitat de Suport a la Recerca de la Catalunya Central, Fundació Institut Universitari per a la Recerca a l'Atenció Primària de Salut Jordi Gol i Gurina, Manresa, Spain, Manresa, Barcelona 08242, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garaulet M, Canteras M, Morales E, Lopez-Guimera G, Sanchez-Carracedo D, Corbalan-Tutau MD. Validation of a questionnaire on emotional eating for use in cases of obesity: the Emotional Eater Questionnaire (EEQ). Nutr Hosp. 2012 Mar-Apr;27(2):645-51. doi: 10.1590/S0212-16112012000200043. PMID 22732995
- [Background] Jeschke N, Nelson PE, Marasas WF. Toxicity to ducklings of Fusarium moniliforme isolated from corn intended for use in poultry feed. Poult Sci. 1987 Oct;66(10):1619-23. doi: 10.3382/ps.0661619. PMID 3432189
- [Background] Garcia-Alvarez A, Serra-Majem L, Ribas-Barba L, Castell C, Foz M, Uauy R, Plasencia A, Salleras L. Obesity and overweight trends in Catalonia, Spain (1992-2003): gender and socio-economic determinants. Public Health Nutr. 2007 Nov;10(11A):1368-78. doi: 10.1017/S1368980007000973. PMID 17988408
- [Background] Ahern AL, Wheeler GM, Aveyard P, Boyland EJ, Halford JCG, Mander AP, Woolston J, Thomson AM, Tsiountsioura M, Cole D, Mead BR, Irvine L, Turner D, Suhrcke M, Pimpin L, Retat L, Jaccard A, Webber L, Cohn SR, Jebb SA. Extended and standard duration weight-loss programme referrals for adults in primary care (WRAP): a randomised controlled trial. Lancet. 2017 Jun 3;389(10085):2214-2225. doi: 10.1016/S0140-6736(17)30647-5. Epub 2017 May 3. PMID 28478041
- [Background] Gomez-Huelgas R, Jansen-Chaparro S, Baca-Osorio AJ, Mancera-Romero J, Tinahones FJ, Bernal-Lopez MR. Effects of a long-term lifestyle intervention program with Mediterranean diet and exercise for the management of patients with metabolic syndrome in a primary care setting. Eur J Intern Med. 2015 Jun;26(5):317-23. doi: 10.1016/j.ejim.2015.04.007. Epub 2015 Apr 20. PMID 25907985
- [Background] Leblanc ES, O'Connor E, Whitlock EP, Patnode CD, Kapka T. Effectiveness of primary care-relevant treatments for obesity in adults: a systematic evidence review for the U.S. Preventive Services Task Force. Ann Intern Med. 2011 Oct 4;155(7):434-47. doi: 10.7326/0003-4819-155-7-201110040-00006. PMID 21969342
- [Background] Paul-Ebhohimhen V, Avenell A. A systematic review of the effectiveness of group versus individual treatments for adult obesity. Obes Facts. 2009;2(1):17-24. doi: 10.1159/000186144. Epub 2009 Feb 3. PMID 20054200
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Jebb SA, Ahern AL, Olson AD, Aston LM, Holzapfel C, Stoll J, Amann-Gassner U, Simpson AE, Fuller NR, Pearson S, Lau NS, Mander AP, Hauner H, Caterson ID. Primary care referral to a commercial provider for weight loss treatment versus standard care: a randomised controlled trial. Lancet. 2011 Oct 22;378(9801):1485-92. doi: 10.1016/S0140-6736(11)61344-5. Epub 2011 Sep 7. PMID 21906798
- [Background] Greaves CJ, Sheppard KE, Abraham C, Hardeman W, Roden M, Evans PH, Schwarz P; IMAGE Study Group. Systematic review of reviews of intervention components associated with increased effectiveness in dietary and physical activity interventions. BMC Public Health. 2011 Feb 18;11:119. doi: 10.1186/1471-2458-11-119. PMID 21333011
- [Background] Salas-Salvado J, Diaz-Lopez A, Ruiz-Canela M, Basora J, Fito M, Corella D, Serra-Majem L, Warnberg J, Romaguera D, Estruch R, Vidal J, Martinez JA, Aros F, Vazquez C, Ros E, Vioque J, Lopez-Miranda J, Bueno-Cavanillas A, Tur JA, Tinahones FJ, Martin V, Lapetra J, Pinto X, Daimiel L, Delgado-Rodriguez M, Matia P, Gomez-Gracia E, Diez-Espino J, Babio N, Castaner O, Sorli JV, Fiol M, Zulet MA, Bullo M, Goday A, Martinez-Gonzalez MA; PREDIMED-Plus investigators. Effect of a Lifestyle Intervention Program With Energy-Restricted Mediterranean Diet and Exercise on Weight Loss and Cardiovascular Risk Factors: One-Year Results of the PREDIMED-Plus Trial. Diabetes Care. 2019 May;42(5):777-788. doi: 10.2337/dc18-0836. Epub 2018 Nov 2. PMID 30389673
- [Background] Gomez Puente JM, Martinez-Marcos M. Overweight and obesity: effectiveness of interventions in adults. Enferm Clin (Engl Ed). 2018 Jan-Feb;28(1):65-74. doi: 10.1016/j.enfcli.2017.06.005. Epub 2017 Dec 21. English, Spanish. PMID 29274691
- [Background] Look AHEAD Research Group; Wadden TA, West DS, Delahanty L, Jakicic J, Rejeski J, Williamson D, Berkowitz RI, Kelley DE, Tomchee C, Hill JO, Kumanyika S. The Look AHEAD study: a description of the lifestyle intervention and the evidence supporting it. Obesity (Silver Spring). 2006 May;14(5):737-52. doi: 10.1038/oby.2006.84. PMID 16855180
- [Background] Appel LJ, Clark JM, Yeh HC, Wang NY, Coughlin JW, Daumit G, Miller ER 3rd, Dalcin A, Jerome GJ, Geller S, Noronha G, Pozefsky T, Charleston J, Reynolds JB, Durkin N, Rubin RR, Louis TA, Brancati FL. Comparative effectiveness of weight-loss interventions in clinical practice. N Engl J Med. 2011 Nov 24;365(21):1959-68. doi: 10.1056/NEJMoa1108660. Epub 2011 Nov 15. PMID 22085317
- [Background] Wharton S, Lau DCW, Vallis M, Sharma AM, Biertho L, Campbell-Scherer D, Adamo K, Alberga A, Bell R, Boule N, Boyling E, Brown J, Calam B, Clarke C, Crowshoe L, Divalentino D, Forhan M, Freedhoff Y, Gagner M, Glazer S, Grand C, Green M, Hahn M, Hawa R, Henderson R, Hong D, Hung P, Janssen I, Jacklin K, Johnson-Stoklossa C, Kemp A, Kirk S, Kuk J, Langlois MF, Lear S, McInnes A, Macklin D, Naji L, Manjoo P, Morin MP, Nerenberg K, Patton I, Pedersen S, Pereira L, Piccinini-Vallis H, Poddar M, Poirier P, Prud'homme D, Salas XR, Rueda-Clausen C, Russell-Mayhew S, Shiau J, Sherifali D, Sievenpiper J, Sockalingam S, Taylor V, Toth E, Twells L, Tytus R, Walji S, Walker L, Wicklum S. Obesity in adults: a clinical practice guideline. CMAJ. 2020 Aug 4;192(31):E875-E891. doi: 10.1503/cmaj.191707. No abstract available. PMID 32753461
- [Background] Rumbo-Rodriguez L, Zaragoza-Marti A, Sanchez-SanSegundo M, Ferrer-Cascales R, Laguna-Perez A, Hurtado-Sanchez JA. Effectiveness of a Two-Year Multicomponent Intervention for the Treatment of Overweight and Obesity in Older People. Nutrients. 2022 Nov 11;14(22):4762. doi: 10.3390/nu14224762. PMID 36432449
- [Background] Lombard CB, Deeks AA, Teede HJ. A systematic review of interventions aimed at the prevention of weight gain in adults. Public Health Nutr. 2009 Nov;12(11):2236-46. doi: 10.1017/S1368980009990577. Epub 2009 Aug 4. PMID 19650959
- [Background] Bluher M. Obesity: global epidemiology and pathogenesis. Nat Rev Endocrinol. 2019 May;15(5):288-298. doi: 10.1038/s41574-019-0176-8. PMID 30814686
- [Background] Gutierrez-Gonzalez E, Garcia-Solano M, Pastor-Barriuso R, Fernandez de Larrea-Baz N, Rollan-Gordo A, Penalver-Argueso B, Pena-Rey I, Pollan M, Perez-Gomez B; ENE-COVID Study Group. Socio-geographical disparities of obesity and excess weight in adults in Spain: insights from the ENE-COVID study. Front Public Health. 2023 Jul 17;11:1195249. doi: 10.3389/fpubh.2023.1195249. eCollection 2023. PMID 37529423
- [Background] Bray GA, Kim KK, Wilding JPH; World Obesity Federation. Obesity: a chronic relapsing progressive disease process. A position statement of the World Obesity Federation. Obes Rev. 2017 Jul;18(7):715-723. doi: 10.1111/obr.12551. Epub 2017 May 10. PMID 28489290
- [Derived] Gargallo-Civil M, Ruiz-Comellas A, Sola L, Vaque-Crusellas C. Energy2MOB study, group food education programme to reduce obesity in adults: randomised clinical trial protocol. BMJ Open. 2025 Dec 21;15(12):e108028. doi: 10.1136/bmjopen-2025-108028. PMID 41423297